CLINICAL TRIAL: NCT06268574
Title: A Multicenter, Open-Label Clinical Trial of RVU120 in Patients With Relapsed or Refractory High-Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia With or Without NPM1 Mutation (RIVER-52)
Brief Title: Safety and Efficacy of RVU120 for Treatment of Relapsed/Refractory AML
Acronym: RIVER-52
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ryvu Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIVER-52
Record Dates: First submitted 2024-01-05; First posted 2024-02-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia (AML); High-risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RVU120 single agent (Experimental): RVU120 oral capsules administered at dose of 250 mg every other day on Days 1-13 of each 21-day cycle of treatment.
  Interventions: Drug: RVU120

INTERVENTIONS:
Drug: RVU120 — RVU120 is a potent, selective inhibitor of CDK8 and its paralog CDK19
  Other Names: SEL120

SUMMARY:
The goal of this study is to assess the safety, tolerability, anti-tumor activity (efficacy), pharmacokinetics (PK), and pharmacodynamics (PD) of the agent RVU120 when administered to adult patients with relapsed or refractory acute myeloid leukemia (AML) or relapsed or progressing high-risk myelodysplastic syndrome (HR-MDS) and who have no alternative therapies available. The study consists of two parts. Part 1 will assess the safety and tolerability of the dosages given and the level of anti-tumor activity or clinical response. Based on the results from part 1 the study will continue to enrol patient into Part 2 which will continue to evaluate safety and tolerability and anti-tumor activity in a larger number of patients.

DETAILED DESCRIPTION:
Patients entering the study will undergo a Screening Period of up to 21 days, a Treatment Period where they will take the drug every other day (7 times in 13 days) in cycles of 21 days, an End of Treatment period (lasting approximately 30 days after last dose), and a 1-year Follow-up Period where participants will be contacted every 3 months for progression and survival status. In Part 1, patients with AML or HR-MDS will be enrolled. All patients will receive RVU120 until the patient meets eligibility for transplant, until there is disease progression or if there are signs of intolerance. A patient may withdraw from the study at any time at their own request or may be withdrawn at any time at the discretion of the Investigator. Depending on the outcome of part 1, part 2 may include patients with HR-MDS and AML irrespective of NPM1 mutation status.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign a written informed consent document and complete study related procedures
* Patients must have a diagnosis of AML or HR-MDS (per 2022 WHO classification) with MDS confirmed as high risk with IPSS-R
* Patients must have relapsed or refractory AML (per ELN 2022 criteria)
* Patients must have relapsed or progressing HR-MDS (per IWG response criteria)
* Patients must have failed first-line treatment and have no alternative therapeutic options likely to produce clinical benefit
* Patients must have ECOG performance status of 0 to 2
* Patients must have adequate end organ function defined as:

  1. WBC < 30 x 10(9)/L on Day 1 prior to first dose of study drug
  2. Platelet count > 10,000/mcL on Day 1 prior to first dose of study drug
  3. Serum albumin ≥ 25 g/L (2.5 g/dL)
  4. Normal coagulation (elevated international normalized ratio [INR], prothrombin time or activated partial thromboplastin time [APTT] <1.3 x the upper limit of normal [ULN] acceptable)
  5. AST (aspartate transaminase) and ALT (alanine transaminase) ≤ 3 x ULN (upper limit of normal)
  6. Total bilirubin ≤ 3 x ULN
  7. Creatinine clearance (Cockcroft & Gault formula) ≥ 30 mL/min

Exclusion Criteria:

* Active central nervous system (CNS) leukemia.
* Diagnosis of acute promyelocytic leukemia (APL), the M3 subtype of AML.
* Previous treatment with CDK8 and/or CDK19-targeted therapy.
* Major surgery within 28 days prior to first dose of study drug.
* Hematopoietic stem cell transplant within 120 days prior to first dose of study drug.
* Active, ≥Grade 2 acute graft versus host disease (GVHD), active moderate-to-severe chronic GVHD, or requirement for systemic immunosuppressive medications for GVHD
* Evidence of ongoing and uncontrolled systemic bacterial, fungal, or viral infection and acute inflammatory conditions (including pancreatitis).
* Known seropositivity or history of active viral infection with human immunodeficiency virus (HIV).
* Ongoing significant liver disease
* Impairment of gastrointestinal function or gastrointestinal disease
* Ongoing drug-induced pneumonitis.
* Concurrent participation in another investigational clinical trial.
* Taking any medications, herbal supplements, or other substances (including smoking) that may interfere with the metabolism of the study drug
* Significant cardiac dysfunction defined as myocardial infarction within 12 months of first dose of study drug, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled dysrhythmias, poorly controlled angina or left ventricular ejection fraction (LVEF) <40% as per echocardiography or multiple gated acquisition (MUGA) scan.
* History of ventricular arrhythmia, or QTc ≥470 ms (Bazett's formula).
* Prior history of malignancies other than AML, unless the participant has been free of the disease for 5 years or more prior to Screening
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR), with and without measurable residual disease (MRD) | 12 months
  Rate of CR, CRh, or CRi

SECONDARY OUTCOMES:
Overall response rate | 12 months
  Overall response rate including CR, CRh, CRi, MLFS, or PR in AML patients or CR, PR, or marrow CR HR-MDS patients
Duration of response | 12 months
  Time from first response to hematologial replase or death
Progression-free survival | 12 months
  Time from first treatment to the first occurrence of disease progression or death
Overall survival | 12 months
  Time from first treatment to death
Incidence of Adverse Events (Safety and Tolerability) | Up to 24 months
  Number and grade of adverse events assessed by CTCAE v5.0
Percentage of participants bridged to hematopoietic stem cell transplantation | 12 months
  Number of hematopoietic stem cell transplantations following response
Maximum Plasma Concentration (Cmax) | 12 months
  Assessment of the peak plasma concentration (Cmax)
Maximum Plasma Concentration (Tmax) | 12 months
  Assessment of the time to peak plasma concentration (Tmax)
Area Under the Concentration Time-Curve (AUC) | 12 months
  Assessed of the area under the plasma concentration versus time curve (AUC)
Impact of treatment on hematological malignancy patient-reported outcomes (HM-PRO) | Up to 12 months
  Assess changes in summary scores of the HM-PRO using a three point impact scale (Not at all, A little, A lot) and a three-point severity scale (Not at all, Mild, Severe)
Impact of treatment on health-related quality of life (QOL-E) | Up to 12 months
  Assess changes in summary scores of the QOL-E questionnaires using a four point scale in order of impact or severity from better to worse outcome (eg, Never, Rarely, Sometimes, Often)

CONTACTS AND LOCATIONS:
Locations (41):
- France (8):
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Universitaire de Lille (CHU Lille), Lille
  - Institut Paoli Calmettes (IPC), Marseille
  - Centre Hospitalier Universitaire (CHU) de Nice - Hopital L'Archet I, Nice
  - Centre Hospitalier Universitaire de Nimes (CHU) - Institut de Cancerologie du Gard, Nîmes
  - Publique-Hopitaux de Paris (AP-HP) - Hopital Saint-Louis, Paris
  - UNICANCER - Centre Henri-Becquerel, Rouen
- Italy (11):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Univerisity of Bologna Policlinico Sant'Orsola, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Careggi University Hospital, Florence
  - Ospedale Vito Fazzi Lecce, Lecce
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST S.r.l., Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata, Roma
  - Humanitas Mirasole S.p.A., Rozzano
  - Azienda Ospedaliera Universitaria Citta Della Salute E Della Scienza Di Torino, Turin
- Poland (12):
  - MTZ Clinical Research, Warsaw, Mazowieckie Województwo
  - Wojewodzki Szpital Specjalistyczny w Bialej Podlaskiej, Biała Podlaska
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii Im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Gliwice
  - Pratia Hematologia Sp. z o.o., Katowice
  - Szpital Wojewodzki Im. Dr. Ludwika Rydygiera w Suwalkach, Suwałki
  - MICS Centrum Medyczne Toruń, Torun
  - Instytut Hematologii I Transfuzjologii, Warsaw
  - Wojskowy Instytut Medyczny Panstwowy Instytut Badawczy, Warsaw
  - Specjalistyczny Szpital Im. Dra Alfreda Sokolowskiego, Wałbrzych
  - Dolnoslaskie Centrum Onkologii Pulmonologii i Hematologii, Wroclaw
  - Szpital Uniwersytecki Imienia Karola Marcinkowskiego w Zielonej Gorze Sp. z o. o., Zielona Góra
- Spain (10):
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Institut Catala d'Oncologia Hospitalet, Barcelona
  - Complejo Hospitalario De Caceres - Hospital General San Pedro De Alcantara, Cáceres
  - Hospital Universitario La Paz (HULP), Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Virgen del Rocío University Hospital, Seville
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No